CLINICAL TRIAL: NCT06602817
Title: The I-gel Plus Supraglottic Airway Device for Elective Surgical Procedures in Prone Position
Brief Title: I-gel Plus Supraglottic Airway Device for Surgical Procedures in Prone Position
Status: Completed | Type: Observational
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Responsible Party: Sponsor
Other Study IDs: 2024-101343-BO-ff
Record Dates: First submitted 2024-09-16; First posted 2024-09-19 (Actual); Last update posted 2025-06-08 (Actual); Status verified 2025-06

CONDITIONS: General Anesthesia; Airway Management; Supraglottic Airway
Keywords: Prone position; Surgery; Airway management

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Surgery in prone position: Patients undergoing elective surgery in prone position with i-gel Plus used for airway management
  Interventions: Other: Exposure: prone position
- Surgery in supine position: Existing prospective control cohort with patients undergoing elective surgery in supine position with i-gel Plus used for airway management
  Interventions: Other: Exposure: Supine position

INTERVENTIONS:
Other: Exposure: prone position — Exposure: surgery in prone position
  Groups: Surgery in prone position
Other: Exposure: Supine position — Exposure: Surgery in supine position
  Groups: Surgery in supine position

SUMMARY:
I-gel Plus is a novel supraglottic airway device that has been evaluated in various studies with high success and low complication rates. Feasibility of supraglottic airway devices (SGA) in patients undergoing surgery in prone position has been demonstrated in some pilot studies and case series; however, the evidence is still limited. It is currently uncertain, if the i-gel Plus facilitates appropriate ventilation in individuals undergoing elective surgery in prone position.

The primary aim of this single-center non-inferior study is to assess the leak fraction of the i-gel Plus in patients undergoing surgery in prone position and to compare it with data from an existing prospective control cohort in patients undergoing surgery in supine position. Secondary aims are to investigate the oropharyngeal seal pressure and other secondary outcome parameters and to compare them with the control cohort.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduling for elective surgery in prone position
* Planned airway management using a SGA
* Adult patients (age 18-89 years)
* ASA physical status 1-3

Exclusion Criteria:

* Pregnant or breastfeeding women
* Non-fasted patients
* Increased risk of aspiration or other contraindications for supraglottic mask ventilation
* Shared airway or intracavity open surgery
* Body mass index (BMI) >35 kg/m2
* Inability to understand or sign informed consent

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients undergoing elective surgery in prone position with i-gel Plus used for airway management
Sampling Method: Non-Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2024-10-01 (Actual); Primary Completion 2025-02-04 (Actual); Study Completion 2025-02-04 (Actual)

PRIMARY OUTCOMES:
Leak fraction | 3 hours
  Ventilation parameter - Leakage volume per tidal volume

SECONDARY OUTCOMES:
Oropharyngeal seal pressure [cm H2O] | 3 hours
  Clinical assessment - leak pressure with audible leak
Leakage volume (ml) | 3 hours
  Ventilation parameter - as displayed on the ventilator
Tidal volume (ml) | 3 hours
  Ventilation parameter - as displayed on the ventilator
Inspiratory peak pressure (cm H2O) | 3 hours
  Ventilation parameter - as displayed on the ventilator
Positive endexpiratory pressure (PEEP) (cm H2O) | 3 hours
  Ventilation parameter - as displayed on the ventilator
Respiratory rate (1/min) | 3 hours
  Ventilation parameter - as displayed on the ventilator
Minute ventilation (l/min/kg) | 3 hours
  Ventilation parameter -as displayed on the ventilator
Endtidal CO2 [mmHg] | 3 hours
  Ventilation parameter - as displayed on the ventilator
Number of insertion attempts | 3 hours
  Clinical assessment - SGA insertion attempts
Insertion success rate (%) | 3 hours
  Clinical assessment
First-attempt insertion success rate (%) | 3 hours
  Clinical assessment - successful placement in only one insertion attempt
Necessity of adjustment maneuvers during the procedure | 3 hours
  Clinical assessment
Insertion time (sec) | 3 hours
  Clinical assessment
Lowest oxygen saturation (%) | 3 hours
  Measured by pulse oximetry
Difficulty of insertion | 3 hours
  Clinical assessment on a scale between 1-5
Ease of gastric tube insertion | 3 hours
  Clinical assessment - rating on a scale from 1-5
Postoperative complications | 24 hours postoperatively
  Clinical assessment
Complications at the end of surgery | 3 hours
  Clinical assessment

CONTACTS AND LOCATIONS:
Overall Officials: Martin Petzoldt, MD, Principal Investigator — University Medical Center Hamburg-Eppendorf: Universitatsklinikum Hamburg-Eppendorf
Locations (1):
- University Medical-Center Hamburg Eppendorf, Hamburg, Hamburg, Germany

IPD SHARING:
Plan to Share IPD: No